CLINICAL TRIAL: NCT02798705
Title: Physiologic Assessment of Microvascular Function in Patients With Cardiac Amyloidosis: Prospective Registry and Pilot Study
Brief Title: Physiologic Assessment of Microvascular Function in Patients With Cardiac Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant professor, Samsung Medical Center
Other Study IDs: AMYL2016-04-122
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Amyloidosis
Keywords: Cardiac amyloidosis; Fractional flow reserve; Microvascular dysfunction; Coronary flow reserve; Index of microcirculatory resistance
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to evaluate coronary flow reserve (CFR), index of microcirculatory resistance (IMR), and proportion of overt microvascular disease, defined as depressed CFR as well as elevated IMR in patients with cardiac amyloidosis. The second objective of this study is to compare results of non-invasive test including serum light chain amount, Doppler echocardiography with 2D strain, and cardiac perfusion MRI. The third object of this study is to evaluate the association between physiologic indices and pathologically measured percent area involvement of interstitium.

DETAILED DESCRIPTION:
Amyloidosis is rare systemic disorder characterized by the extracellular deposition of misfolded protein in various organ system, including heart. Among the several types of amyloid fibrils, the light chain and transthyretin amyloid proteins most commonly affect the heart.

Cardiac amyloid deposits result in increased ventricular wall thickness and produce a restrictive cardiomyopathy presenting primarily as biventricular congestive heart failure. Anginal symptoms and signs of ischemia have been reported in some patients with cardiac amyloidosis without obstructive epicardial coronary artery disease (CAD). Autopsy studies have shown amyloid deposits around and between cardiac myocytes in the interstitium, the perivascular regions, and the media of intramyocardial coronary vessels. Amyloidosis is thus a prime example of a disorder with the potential to cause coronary microvascular dysfunction via 3 major mechanisms: (1) structural (amyloid deposition in the vessel wall causing wall thickening and luminal stenosis), (2) extravascular (extrinsic compression of the microvasculature from perivascular and interstitial amyloid deposits and decreased diastolic perfusion), and (3) functional (autonomic and endothelial dysfunction).

Previous basic research presented that adipose arteriole or atrial coronary arterioles showed endothelial dysfunction even after brief exposure to physiologic amounts of light chain, and also showed increased oxidative stress, reduced NO bioavailability, and peroxynitrite production. All these previous evidences imply that coronary microvascular dysfunction and subsequent global ischemic insult can be precursor of overt diastolic or systolic dysfunction in patients with cardiac amyloidosis.

However, there have only 1 study which evaluated microvascular function in vivo using N13-ammonium positron emission tomography (PET). In that study, Dorbala et al. demonstrated that amyloidosis patients showed depressed global resting myocardial blood flow (MBF), stress MBF, and CFR and higher minimal coronary vascular resistance, compared with patients with left ventricular hypertrophy. However, low availability, high cost, and limited resolution of N13 ammonium PET precludes the generalizability of the results.

Since thermodilution-derived coronary flow reserve and index or microcirculatory reserve using pressure-temperature wire has been well validated prognostic index in assessment of patients with coronary artery disease or functionally insignificant epicardial coronary stenosis, invasive physiologic assessment might more specifically assess macro- and microvascular function in patients with cardiac amyloidosis. Moreover, adding physiologic measurement in the current frame in diagnosis of cardiac amyloidosis might enhance risk stratification of patients.

Therefore, the current study will perform physiologic assessment including fractional flow reserve, coronary flow reserve, and index of microcirculatory resistance in patients with cardiac amyloidosis, and explore correlation among the physiologic indices and conventional measurements of echocardiography, perfusion MRI, serum light chain amount, or NT-proBNP. In addition, the differences of physiologic indices according to disease severity of cardiac amyloidosis, which measured by endomyocardial biopsy findings will be also explored. Since there was no previous study which performed invasive physiologic assessment in amyloidosis patients, this study will be performed as pilot study. Target sample size will be at least 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject age 18-85 years old
* Patients with confirmed cardiac amyloidosis by heart biopsy
* Patients with confirmed amyloidosis by biopsy other than heart and evidence of cardiac involvement in echocardiography
* Patients who underwent invasive physiologic assessment within 3 months from diagnosis of primary disease

Exclusion Criteria:

* Patients with cardiogenic shock
* Patients with unstable vital sign that precludes coronary angiography
* Patients with major bleeding in last 3 months
* Patients with active bleeding
* Patients with coagulopathy
* Patients with severe valvular heart disease
* Patients who refused to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically confirmed amyloidosis patients with suspected cardiac involvement undergoing coronary angiography for coronary disease evaluation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-04-11 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 2 Years
  Comparison of all-cause mortality in amyloidosis patients with or without microvascular disease

SECONDARY OUTCOMES:
Correlation between IMR and echocardiographic parameters | within 3 months of diagnosis
  Correlation between IMR and echocardiographic parameters (E/E', LV ejection fraction, etc.)
Correlation between IMR and serum biochemicalmarkers | within 3 months of diagnosis
  Correlation between IMR and serum biochemicalmarkers (troponin T, NT-proBNP, serum free light chain)
Distribution of CFR or IMR according to pathologic severity of myocardial involvement | within 3 months of diagnosis
  Distribution of CFR or IMR according to pathologic severity of myocardial involvement (Percent amyloid load)
Comparison of CFR or IMR value in amyloidosis patient with or without relative perfusion defect in myocardial perfusion imaging (ex> adenosine-SPECT or perfusion MRI) | within 3 months of diagnosis
Comparison of CFR or IMR value in different type of amyloidosis (AL type, hereditary type, AA type, senile type) | within 3 months of diagnosis
Comparison of CFR or IMR value in amyloidosis patient according to current staging by Troponin T, NT-proBNP and free light chain difference | within 3 months of diagnosis
Optimal cut-off values of physiologic indices (CFR, IMR) for prediction of all-cause mortality | 2 Years
Association between physiologic indices and pathologically measured percent area involvement in myocardial interstitium | within 3 months of diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center; Eun-Seok Jeon, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked

REFERENCES:
- [Derived] Choi KH, Lee JM, Kim SR, Kim D, Choi JO, Kim SJ, Kim K, Kim JS, Koo BK, Jeon ES. Prognostic Value of the Index of Microcirculatory Resistance Over Serum Biomarkers in Cardiac Amyloidosis. J Am Coll Cardiol. 2020 Feb 11;75(5):560-561. doi: 10.1016/j.jacc.2019.11.045. No abstract available. PMID 32029139